CLINICAL TRIAL: NCT05520216
Title: Effect of Rib Cage and Spine Mobility on Maximum Breath-Hold Time
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: Thesis; 21/778 (Other: Sağlık Bilimleri University)
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-07

CONDITIONS: Healthy Participant
Keywords: Maximum breath hold test; Spinal Mouse; Mobility
MeSH Terms: interventions — 4-Acetamido-4'-isothiocyanatostilbene-2,2'-disulfonic Acid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- asymptomatic individuals: The demographic information of the participants (gender, age, height, body weight, body mass index, occupation, dominant extremity, education level, marital status) will be questioned with the Demographic Data Form to be created by the researchers. Except for the demographic data form, the breath-holding capacity of the participants will be evaluated by measuring the breath-holding times, and the thoracic cage mobility will be evaluated by measuring the chest circumference during normal respiration, maximal inspiration and maximal expiration. The curvature of the spine, the presence of kyphosis and lordosis will be measured using the Spinal Mouse (IDIAG m360) device, which is an objective measurement method. The flexibility of the spine and indirectly the mobility of the rib cage will be checked with the sit and lie test. The results of the evaluations will be recorded.
  Interventions: Device: Spinal mouse (idiag m360); Behavioral: chest circumference measurement; Behavioral: Maximum Breath Hold Test; Behavioral: Sit and Reach

INTERVENTIONS:
Device: Spinal mouse (idiag m360) — A noninvasive Spinal Mouse device will be used to measure the thoracic kyphosis and lumbar lordosis angle of the spinal column in the sagittal plane. It will be displayed on the computer aided software screen where the thoracic and lumbar region angles are calculated by swiping over the spinal processes from top to bottom with the Spinal Mouse (IDIAG m360) device. Measurements will be taken while standing on a flat surface. The volunteer will take off his upper clothes and shoes during the examination. Relax your arms and torso will be positioned next to you. The distance between the feet will be approximately waist width and parallel to each other, the knees will be straight and face motionless. He will stand where he feels comfortable. A Spinal Mouse examination will be performed and data will be recorded.
Behavioral: chest circumference measurement — Measurements will be taken from the axillary (4th rib level - two fingers below the axilla), epigastric (xiphoid process level) and subcostal (9th rib level) regions at the time of normal, maximal inspiration, and maximal expiration using a tape measure while the patient is in a sitting position. The tape measure will be placed in the area to be measured. Care will be taken that there is no folding or horizontal level difference in the tape measure and that the fingers are not under the tape measure. Normal respiration will be measured first and recorded in centimeters (cm). The patient will then be asked to take a deep, long breath towards the bottom of the tape measure. The value obtained will be recorded as the deep inspiration value. Immediately after deep inspiration, the patient will be asked to make a deep and long expiration. The obtained value will be recorded as deep expiration.
Behavioral: Maximum Breath Hold Test — During the breath-hold measurement, the subject will sit in a chair with a backrest. He will take a deep breath through his nose. We do not want maneuvers (Valsalva and Müller) and diaphragm contractions that will affect the breath-hold time, so volunteers will be observed throughout the test. The test will be terminated as soon as involuntary diaphragm contractions are seen. This test will be applied 3 times by resting the volunteer with breaks for 5 minutes. The average of 3 test results will be taken (Lin, Y. C.: Effect of O2 and CO2 on breath hold breaking point. In The Physiology of Breath Hold Diving. (eds): CEG Lundgren, M Ferringo, Undersea and Hyperbaric Medical Society Inc, Bethesda, Maryland, p: 75-87 1987.).
Behavioral: Sit and Reach — While the participant is sitting on the floor with his back to the wall and his legs are fully extended in front of him, his knees should be in full contact with the floor. The box will be placed on the sole of the participant's feet (without shoes) in full contact with the volunteer's feet. The participant will be instructed to lean forward as slowly as possible, keeping their fingertips level with each other and their legs straight on the floor. He will be asked to slowly lie down along the ruler three times, and on the third attempt the volunteer will be instructed to reach out as far as possible and hold for 2 seconds. This value will be saved

SUMMARY:
In this study, it was aimed to look at the effect of rib cage and spine mobility on maximum breath holding time. To determine the relationship between spine and rib cage mobility level and respiratory capacity.

DETAILED DESCRIPTION:
The demographic information of the participants (gender, age, height, body weight, body mass index, occupation, dominant extremity, education level, marital status) will be questioned with the Demographic Data Form to be created by the researchers. Except for the demographic data form, the breath-holding capacity of the participants will be evaluated by measuring the breath-holding times, and the thoracic cage mobility will be evaluated by measuring the chest circumference during normal respiration, maximal inspiration and maximal expiration. The curvature of the spine, the presence of kyphosis and lordosis will be measured using the Spinal Mouse (IDIAG m360) device, which is an objective measurement method. The flexibility of the spine and indirectly the mobility of the rib cage will be checked with the sit and lie test. The results of the evaluations will be recorded.

A consent form stating that they are healthy female and male volunteer participants aged between 18-25 years old and who meet the inclusion criteria will be filled in to participate in the study. After the consent form is signed, clinical evaluations will begin.

Study Design: Experimental nonrandomized field study

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-25
* Being cooperative
* Those who want to participate in the study voluntarily

Exclusion Criteria:

* Having had any lower extremity or spine surgery
* Having a vestibular system disorder
* Pregnancy or the possibility of pregnancy
* Known, diagnosed spinal cord, visceral, or other musculoskeletal disorders
* Refusal to participate in the study

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: asymptomatic individual
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2022-09-20 (Estimated); Primary Completion 2023-01-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Maximum breat-hold time | 20 05 2022
  In conclusion, in this study, a significant relationship was found between maximum breath holding time and age, BMI, and smoking.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu DEMİR, Principal Investigator — Saglik Bilimleri University
Locations (1):
- Saglik Bilimleri University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Masaki M, Ogawa Y, Inagaki Y, Sato Y, Yokota M, Maruyama S, Takeuchi M, Kasahara M, Minakawa K, Okamoto M, Chiyoda Y, Mino K, Aoyama K, Nishi T, Ando Y. Association of sagittal spinal alignment in the sitting position with the trunk and lower extremity muscle masses in children and adults with cerebral palsy: A pilot study. Clin Biomech (Bristol). 2021 Dec;90:105491. doi: 10.1016/j.clinbiomech.2021.105491. Epub 2021 Sep 25. PMID 34597916